CLINICAL TRIAL: NCT00313365
Title: Arthrotomy With Irrigation and Debridement Versus Serial Arthrocentesis as Treatment for Septic Arthritis in Adults
Brief Title: Surgical Lavage vs Serial Needle Aspiration for Infected Joints
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never started because Dr. Hammerberg left before it could be started.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas Moore, Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218-2006
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Arthritis; Septic
MeSH Terms: conditions — Arthritis | interventions — Arthrocentesis

INTERVENTIONS:
Procedure: Surgical Lavage (Arthrotomy)
Procedure: Arthrocentesis (Serial needle aspiration)

SUMMARY:
Joint spaces are aseptic areas, meaning that they do not contain microorganisms. Any injury to the joint space could cause the entry of microorganisms, with the potential to cause infection. Septic arthritis refers to the infection of a joint space with microorganisms, usually bacteria. This invasion initiates a process of inflammation and causes irreversible damage to a joint cavity. Patients typically present with pain, swelling, decreased motion, and inability to use the joint. When bacteria enter a joint space, the host immune system responds by concentrating inflammatory cells within the joint. While inflammatory cells serve to eliminate the bacteria, they also produce substances that not only attack bacteria but also could destroy the joint space. These substances are called enzymes, and they could damage the cartilage (translucent fairly elastic tissue around the joint) and adjacent bone in the process. Because cartilage has a poor ability to cure itself, this process may lead to irreversible damage and chronic joint dysfunction. Studies have found that signs of early joint damage can be found within hours following joint infection. This is true even if antibiotic therapy (medicine to fight the infection) is started within 24 hours of infection. Also, delay in treatment has been related to poor outcome. However, the best method of treating septic arthritis has yet to be determined. Currently, there are two accepted ways for treating septic arthritis: serial needle aspiration (introducing a needle in the joint to aspirate the inflammatory liquid), and surgical lavage (opening and cleaning the joint space in the OR under anesthesia). Antibiotics are also used with these two forms of treatment. Supporters of surgery believe that the most dependable method of eliminating bacteria from a joint space is through arthrotomy (opening the joint with a surgical incision) and lavage (irrigation of the joint with copious saline solution) .Promoters of serial needle aspiration support this method because it is quick, does not require opening the joint space, and can be performed without anesthesia.At present, there are no conclusive studies comparing the two techniques. Hopefully, this study will help delineate the best course of management.

DETAILED DESCRIPTION:
The principle objectives and justification for this study:

To determine whether arthrotomy with irrigation and debridement or repeated arthrocentesis provides a clear benefit over the other for the treatment of septic arthritis in adults.

Background:

Septic arthritis is an infection with consequential inflammation of a joint space by various microorganisms. Typically it is bacterial in origin and results by hematological seeding or direct invasion of a joint space. This invasion initiates a cascade of inflammation and causes irreversible damage to a joint cavity. Patients typically present with edema, erythema, substantial decrease in range of motion, and the inability to use the joint. It remains a significant medical issue accounting for 0.2-0.7% of hospital admissions in the United States with a mortality rate ranging from 2-14%.

Once bacteria enter a joint space it produces a purulent fluid that induces an acute inflammatory response. The body's inflammatory cells, although aids in eradicating the bacteria, produces enzymes that also damage extracellular cartilage matrix, synovium, and adjacent bone in a relatively short period of time.1,2 Because adult cartilage has poor regenerative capabilities, this process leads to irreversible damage and chronic joint dysfunction.4 Studies have found that signs of early joint damage can be found within hours following joint infection.1, 5 This is true even if antibiotic therapy is started within 24 hours of infection. Also, delay in initiation of treatment has repeatedly found to be a major determinant of poor outcome.6 Thus, it is well accepted that early drainage of purulent material in addition to antibiotics is imperative for preventing irreparable articular damage.4 However, the best method for doing so has yet to be determined.

Currently studies have yet to clearly provide an ideal method of management. Although animal models seem to support early surgical intervention, retrospective studies in human reveal that arthrocentesis may provide better outcomes but with an increased risk of mortality.4,7,10 Proponents of surgery believe the proper visualization, debridement, and lavage can only be conducted through surgery thus protecting the articular cartilage from rapid destruction.8-10,12,13 Whereas proponents of medical management argue the needle aspiration is quick, less invasive, and can be conducted multiple times to prevent accumulation of pus and follow effectiveness of antibiotic treatment.7,11

Study Design: Randomized Prospective study.

Selection of Patients: We will select 200 patients admitted to Grady for septic arthritis of the ankle, knee, hip, wrist, elbow, or shoulder.

Inclusion criteria:

* Patients with acute onset of symptoms of less than or equal to two weeks' duration.
* Patients with infection of only the following joints: ankle, knee, hip, wrist, elbow, or shoulder
* Patients with proven bacterial infection by positive gram stain or culture of synovial fluid and with white blood cell count in synovial flood consistent with infection (75,000 - 150,000 cells/mm3.)
* Cases with negative synovial fluid cultures if positive blood cultures are present and associated with typical inflammatory synovial fluid changes without other identifiable sources of infection and if antibiotic therapy had been initiated earlier to explain negative synovial fluid cultures.
* Monoarticular arthritis

Exclusion criteria

* Gonococcal infections
* Infected prosthetic joints
* Adjacent osteomyelitis preceding joint infection
* Septic arthritis occurring as an incidental event late in the course of otherwise fatal illness
* Patients that are 17 years old or less.
* Polyarticular arthritis.

Methods:

Definitive diagnosis for septic arthritis will be made following analysis of the joint fluid for a positive gram stain/culture and white blood cell (WBC) count consistent with infection (75,000-150,000 cells/mm3) as discussed above. Plain films of the involved joint will be acquired to evaluate for soft tissue edema, osteomyelitis, as well as to rule out other pathological involvement. Patients' blood sample will also be evaluated for central blood count (CBC), erythrocyte sedimentation rate (ESR), C- reactive protein (CRP), and cultures.

After the patients are admitted for treatment of the infected joint, they will be asked to participate in the study. The nature of the study will be explained by a member of the orthopaedic department, and signed consent will be obtained prior to inclusion in the study.

Method of Randomization:

There will be two indistinguishable sealed envelopes created at the beginning of the study for each patient enrolled. Inside one envelope will be a piece of paper with Group I written on it. Inside the other envelope will be a piece of paper with Group II written on it. Patients will be randomly placed in either group I receiving arthrotomy with irrigation and debridement or group II undergoing repeated arthrocentesis based upon which envelope is chosen.

Treatment Method for Group I:

Patients undergoing surgical treatment will undergo surgery in the first 72 hours. During the procedure, there will be direct visualization of joint cavity, thorough debridement of any adhesions or necrotic tissue, and irrigation-drainage with saline solution to eliminate as much debris as possible. Synovectomy will not be performed. Temporary drainage catheters will then be inserted into the joint for 48 hours.

Treatment Method for Group II:

The second group will undergo daily bedside arthrocentesis. The involved joint will be prepped and draped in a sterile fashion prior to every aspiration. As much infected joint fluid will be removed as possible. Each aspirated fluid will be evaluated for gross appearance, cell count, gram stain and culture, glucose concentration, and crystal analysis. Arthrocentesis will be performed daily until effusion resolves or until aspirate no longer yields a purulent exudate.

After Treatment Method:

Appropriate antibiotics will be provided to both groups intravenously then changed to oral pills upon discharge for a total course of 14 days following irrigation and debridement or final arthrocentesis. Also physical therapy and pain medications will be provided to all patients. The affected joint will be initially immobilized in a position of function. One the infection is under control, range of motion will be initiated slowly but deliberately.

Laboratory Findings:

Patients' blood sample will also be evaluated and followed for central blood count (CBC), erythrocyte sedimentation rate (ESR), and c-reactive protein (CRP) once daily during hospital stay and once at each follow up appointment.

Method of Follow up:

Patients will be followed up at 2 weeks, 2 months, and 6 months post discharge. At each follow-up appointment, patients will be evaluated for symptomatic improvement as well as examined for residual edema, range of motion, recurrence of infection, radiological changes, and erythema.

Sample size calculation:

A sample size of 100 patients per group achieves 94% statistical power to detect a difference of 20% between the null hypothesis that 90% in both the surgery and aspiration groups will clear infection within 2 months and the alternative hypothesis that the proportion in the aspiration group that clear infection is 70% using a two-sided Z test with continuity correction and unpooled variance (significance level of 0.05). All power calculations were performed with PASS 2005 software. This calculation was performed by Kirk Easley, Senior Associate at the Biostatistics Department, Rollins School of Public Health.

Outcome Measures:

Outcome will be divided into four groups:

Good: if the patient recovered completely without any decrease in range of motion and only experienced minimal residual pain.

Fair: if there is decrease in ROM up to 10%, moderate pain, signs of recurrence Poor: if there is greater than 10% decrease in ROM, >10 degrees of flexion deformity, ankylosis, osteomyelitis, persistent effusion, and/or severe or disabling pain.

Death: Patients who died for any reason in the course of their joint infection

End points for this study would be the absence of infection or the need to have an additional procedure for infection control (i.e. secondary surgical lavage).

Short Form-36 (SF-36), Musculoskeletal Functional Assessment (MFA), and Western Ontario and McMaster Osteoarthritis Index (WOMAC) questionnaires will also be used to assess outcome at each follow-up appointment. The data will be collected into an Excel spreadsheet and analyzed to determine one treatment options significantly improves outcome over the other. Statistical analysis will be achieved by using Fisher's exact test. A P value <0.05 will be considered as statistically significant. This study is not expected to cause any additional risk for our patients because both forms of treatment are accepted as standard of treatment and used nationally.

References:

1. Pioro M, Mandell B. Septic Arthritis. Rheum Dis Clin North Am. 1997; 23:239-257.
2. Donatto K. Orthopedic management of pyogenic arthritis. Comp Ther. 1999;25:411-417.
3. Weston VC, Jones AC, Bradbury N, et al. Clinical features and outcome of septic arthritis in a single UK health district 1982-1991. Ann Rheum Dis. 1999; 58: 214-219.
4. Manadan A, Block J. Daily Needle Aspiration Versus Surgical Lavage for the Treatment of Bacterial Septic Arthritis in Adults. American Journal of Therapeutics 2004. 11, 412-415.
5. Smith LR, Merchant TC, Schurman DL: In vitro cartilage degradation by E. coli and S. aureus. Arthritis Rheum 25:441, 1992
6. Smith JW: Infectious arthritis. Infect Dis Clin North Am 4:523, 1990.
7. Broy SB, Stulberg SD, Schmid F. The role of arthroscopy in the diagnosis and management of the septic joint. Clin Rheum Dis. 1986;12:489-500.
8. Smith RL, Schurman DJ. Comparison of cartilage destruction between infectious and adjuvant arthritis. J Orthop Res. 1983; 1:136-143.
9. Daniel D, Akeson W, Amiel D, et al. Lavage of septic joints in rabbits: effects of chondrolysis. J Bone Joint Surg. 1976; 58: 393-395.
10. Goldstein W, Gleason T, Barmada R. A comparison between arthrotomy and irrigation and multiple aspirations in the treatment of pyogenic arthritis: a histological study in a rabbit model. Orthopedics. 1983;6:1309-1314.
11. Goldenberg D, Brandt K, Cohen A, et al. Treatment of septic arthritis: comparison of needle aspiration and surgery as initial modes of joint drainage. Arthritis Rheum. 1975; 18:83-90.
12. Parisen J, Shaffer B. Arthroscopic management of pyarthrosis. Clin Orthop. 1992;275:243-247.
13. Bynum DR, Nunley JA, Goldner JL, et al. Pyogenic arthritis: emphasis on the need for surgical drainage of the infected joint. South Med J. 1982;75:1232.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute onset of symptoms of less than or equal to two weeks' duration.
* Patients with infection of only the following joints: ankle, knee, hip, wrist, elbow, or shoulder
* Patients with proven bacterial infection by positive gram stain or culture of synovial fluid and with white blood cell count in synovial flood consistent with infection (75,000 - 150,000 cells/mm3.)
* Cases with negative synovial fluid cultures if positive blood cultures are present and associated with typical inflammatory synovial fluid changes without other identifiable sources of infection and if antibiotic therapy had been initiated earlier to explain negative synovial fluid cultures.
* Monoarticular arthritis

Exclusion Criteria:

* Gonococcal infections
* Infected prosthetic joints
* Adjacent osteomyelitis preceding joint infection
* Septic arthritis occurring as an incidental event late in the course of otherwise fatal illness
* Patients that are 17 years old or less.
* Polyarticular arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Eradication of infection at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Erick M Hammerberg, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States